CLINICAL TRIAL: NCT02944006
Title: Establishment of Radiomics Database by Clinical Application of Multiparametric MRI Including DCE-MRI Based on Incoherent Undersampling
Brief Title: Establishment of Radiomics Database by Clinical Application of Multiparametric MRI Based on Incoherent Undersampling
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Other Study IDs: 2015-1160
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Pancreas Cancer
Keywords: MRI
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: multi-parametric MRI — multiparametric MRI is performed in all patients, and the sequence includes dynamic contrast enhanced (DCE) MRI, diffusion weighted imaging (DWI), tissue maps, and MR cholangiography.

SUMMARY:
This study aims to establish radiomics database for pancreas cancer from multiparametric MRI including DCE-MRI obtained by using incoherent undersampling and radial acquisition for clinical staging as well as quantitative analysis.

ELIGIBILITY:
Inclusion Criteria:

* surgical candidate for pancreatico-duodenectomy
* characteristic finding of pancreatic adenocarcinoma on prior CT or MRI
* OR histologically diagnosed with pancreatic adenocarcinoma
* signed for informed consent

Exclusion Criteria:

* under 18 years
* not eligible for pancreatico-duodenectomy
* unresectable patients (locally advanced on prior CT/MRI or metastatic disease)
* tumors with suspicion of other histologic types (neuroendocrine, IPMN, etc)
* any contra-indication of contrast-enhanced MRI
* recurred pancreatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to undergo pancreatobiliary MRI as a preoperative workup for suspected resectable pancreas cancer (adenocarcinoma)
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
T-staging | 4 weeks after MR acquisition
  T-staging of the tumor at MRI.

SECONDARY OUTCOMES:
N-staging | 4 weeks after MR acquisition
  N-staging of the tumor at MRI
arterial blood flow | 4 weeks after MR acquisition
  arterial blood flow of the tumor and adjacent parenchma on DCE-MRI
arterial fraction | 4 weeks after MR acquisition
  arterial fraction of the tumor and adjacent parenchyma on DCE-MRI
mean transit time | 4 weeks after MR acquisition
  mean transit time of the tumor and adjacent parenchyma on DCE-MRI
extracellular volume | 4 weeks after MR acquisition
  extracellular volume of the tumor and adjacent parenchyma on DCE-MRI
true diffusion | 4 weeks after MR acquisition
  true diffusion of the tumor and adjacent parenchyma on DWI with intravoxel incoherent motion model
pseudodiffusion | 4 weeks after MR acquisition
  pseudodiffusion of the tumor and adjacent parenchyma on DWI with intravoxel incoherent motion model
perfusion fraction | 4 weeks after MR acquisition
  perfusion fraction of the tumor and adjacent parenchyma on DWI with intravoxel incoherent motion model
kurtosis | 4 weeks after MR acquisition
  kurtosis of the tumor and adjacent parenchyma on DWI with kurtosis model
mean diffusivity | 4 weeks after MR acquisition
  mean diffusivity of the tumor and adjacent parenchyma on DWI with kurtosis model

OTHER OUTCOMES:
T1 value | 4 weeks after MR acquisition
  T1 value of the tumor and adjacent parenchyma using T1 map
T2 value | 4 weeks after MR acquisition
  T1 value of the tumor and adjacent parenchyma using T2 map
fat fraction | 4 weeks after MR acquisition
  fat fraction of the tumor and adjacent parenchyma using T2* corrected fat map
global textural feature | 4 weeks after MR acquisition
  first order parameters related to the grey level frequency distribution in the region of interest using dedicated software
local textural feature | 4 weeks after MR acquisition
  second order parameters calculated with spatial grey level dependence matrices or co-occurrence matrices using dedicated software
attenuation | 4 weeks after MR acquisition
  hounsefield unit (HU) of the tumor and parameter on CT within 4 weeks of MRI
transient dyspnea | 1 day after MR acquisition
  development of transient dyspnea or involuntary motion after contrast media administration

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No